CLINICAL TRIAL: NCT07275619
Title: Normative Data for Cardiorespiratory Fitness in Healthy Adults Using the Queen's College Step Test
Brief Title: Normative Data for Cardiorespiratory Fitness in Healthy Adults
Acronym: NDFCFIHAUTQCST
Status: Enrolling by invitation | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Wajeeha Zia, Assistant Professor, Riphah International University
Other Study IDs: nida naz
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adults
Keywords: Adults; Cardiorespiratory fitness; Normative; Queen's college step test; VO2max

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: 18 - 29 years: Cohort 1 will be approximately 200 consist of 100 males and 100 females. Subjects will be divided into cohort group according to their age. Queen's college step test will be used to estimate the VO2max
- Cohort 2: 30 - 41 years: Cohort 2 will be approximately 200 consist of 100 males and 100 females. Subjects will be divided into cohort group according to their age. Queen's college step test will be used to estimate the VO2max
- Cohort 3: 42 - 53 years: Cohort 3 will be approximately 200 consist of 100 males and 100 females. Subjects will be divided into cohort group according to their age. Queen's college step test will be used to estimate the VO2max
- Cohort 4: 54 - 65 years: Cohort 4 will be approximately 200 consist of 100 males and 100 females. Subjects will be divided into cohort group according to their age. Queen's college step test will be used to estimate the VO2max

SUMMARY:
Cardiorespiratory fitness (CRF) is a physical attribute which represents how effectively various bodily systems work together to transport and utilize oxygen to support muscular activity during prolonged, rhythmic, large-muscle, whole-body exercise. A key element associated with physical fitness is VO2max, which is referred to as cardiorespiratory fitness. Queen's college step test will be used to estimate the VO2max. This study will be cross sectional, normative study. Healthy adults aged 18-65 years from community setting will be recruited through non probability convenient sampling technique to collect data as per inclusion criteria. Sample size will be approximately 800, consist of equal ratio of males and females. Heart Rate, Recovery Heart Rate, VO2 max and METS will be calculated of each subject. Following equation is used to calculate VO2max, for females: VO2max = 65.81- [0.1847× HR] for males: VO2max = 111.33- [0.42× HR]. Data analysis will be conducted by using SPSS (Statistical Package for the Social Sciences) version 28.

DETAILED DESCRIPTION:
Cardiorespiratory fitness (CRF) is a physical attribute which represents how effectively various bodily systems work together to transport and utilize oxygen to support muscular activity during prolonged, rhythmic, large-muscle, whole-body exercise. A key element associated with physical fitness is VO2max, which is referred to as cardiorespiratory fitness. Queen's college step test (reliability = 0.92, validity = 0.75) will be used to estimate the VO2max. The objectives of the study is to obtain the normative reference values for cardiorespiratory fitness in healthy pakistani adults.

This study will be cross sectional, normative study. Healthy adults aged 18-65 years from community setting will be recruited through non probability convenient sampling technique to collect data as per inclusion criteria. Sample size will be approximately 800, consist of equal ratio of males and females. Heart Rate, Recovery Heart Rate, VO2 max and METS will be calculated of each subject. Following equation is used to calculate VO2max, for females: VO2max = 65.81- [0.1847× HR] for males: VO2max = 111.33- [0.42× HR]. Demographics include Age (years), Height (m2), Weight (kg) and Body Mass Index (BMI kg/m2) will be measure for each subject.Data analysis will be conducted by using SPSS (Statistical Package for the Social Sciences) version 28.

Key words:

Adults, Cardiorespiratory fitness, Normative, Queen's college step test, VO2max

ELIGIBILITY:
Inclusion Criteria:

* • Pakistani Adults of age group 18-65 according to ACSM's guidelines

  * Current healthy adults recruited by filling PAR_Q test
  * IPAQ short form will be administered, Participants scoring moderate or high activity level will be selected to perform QCST
  * BMI ≥ 18.5 kg/m2 - ≤ 24.9 kg/m2
  * Resting spO2 >95%
  * Resting heart rate ≥60bpm and ≤100bpm
  * Mentally and physically fit adults without any physical, physiological and psychological issues

Exclusion Criteria:

Presence of any acute/chronic illness Any cardiovascular, respiratory, neuromuscular, psychological, musculoskeletal or orthopedic condition and history of surgery Individuals taking any medical treatment History of active smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Queen's college step test | one time point
  QCST will be used to estimate the VO2max. The step test will be performed using a tool of 16.25 inches height. Stepping will be performed for a total duration of 3 minutes at the rate of 22 steps per minute for females and 24 steps per minute for males which will be set by a metronome. After completing the stepping , the subject remains standing, wait 5 seconds, take a 15s heart rate count and multiply the HR by 4 to convert into beats per minute. following equation is used to predict VO2max.
  For females: VO2max = 65.81- [0.1847× HR] For males: VO2max = 111.33- [0.42× HR] The reliability and validity of queen's college step test is 0.92 and 0.75 respectively.
pulse oximeter | one time point
  Heart rate will be calculated by pulse oximeter. After completing the stepping , the subject remains standing, wait 5 seconds, take a 15s heart rate count and multiply the HR by 4 to convert into beats per minute.
Recovery Heart Rate | one time point
  Recovery heart rate will be measure by substracting the heart rate after 1 minute from the peak heart rate which will be compare with standard values to check the heart health.
METS | one time point
  Metabolic equivalents of task (METS) will be calculated dividing VO2max by 3.5ml/kg/min.
  METS = VO2 MAX ÷ 3.5 ml/kg/min

SECONDARY OUTCOMES:
stadiometer | one time point
  height (m2) will be measure through stadiometer
weighing machine | one time point
  weight (kg) will be measure through weighing machine
Body Mass Index | one time point
  BMI will be calculated dividing weight by height (m2).

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah International University, Lahore, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Kunutsor SK, Isiozor NM, Myers J, Seidu S, Khunti K, Laukkanen JA. Baseline and usual cardiorespiratory fitness and the risk of chronic kidney disease: A prospective study and meta-analysis of published observational cohort studies. Geroscience. 2023 Jun;45(3):1761-1774. doi: 10.1007/s11357-023-00727-3. Epub 2023 Jan 17. PMID 36646903
- [Background] Rossi Neto JM, Tebexreni AS, Alves ANF, Smanio PEP, de Abreu FB, Thomazi MC, Nishio PA, Cuninghant IA. Cardiorespiratory fitness data from 18,189 participants who underwent treadmill cardiopulmonary exercise testing in a Brazilian population. PLoS One. 2019 Jan 9;14(1):e0209897. doi: 10.1371/journal.pone.0209897. eCollection 2019. PMID 30625200
- [Background] Kaminsky LA, Arena R, Myers J. Reference Standards for Cardiorespiratory Fitness Measured With Cardiopulmonary Exercise Testing: Data From the Fitness Registry and the Importance of Exercise National Database. Mayo Clin Proc. 2015 Nov;90(11):1515-23. doi: 10.1016/j.mayocp.2015.07.026. Epub 2015 Oct 5. PMID 26455884
- [Background] Ekblom-Bak E, Ekblom O, Andersson G, Wallin P, Soderling J, Hemmingsson E, Ekblom B. Decline in cardiorespiratory fitness in the Swedish working force between 1995 and 2017. Scand J Med Sci Sports. 2019 Feb;29(2):232-239. doi: 10.1111/sms.13328. Epub 2018 Nov 15. PMID 30351472
- [Background] Hills AP, Jayasinghe S, Arena R, Byrne NM. Global status of cardiorespiratory fitness and physical activity - Are we improving or getting worse? Prog Cardiovasc Dis. 2024 Mar-Apr;83:16-22. doi: 10.1016/j.pcad.2024.02.008. Epub 2024 Feb 27. PMID 38417767
- [Background] Sloan RA. Estimated Cardiorespiratory Fitness and Metabolic Risks. Int J Environ Res Public Health. 2024 May 16;21(5):635. doi: 10.3390/ijerph21050635. PMID 38791849
- [Background] Dourado VZ, Nishiaka RK, Simoes MSMP, Lauria VT, Tanni SE, Godoy I, Gagliardi ART, Romiti M, Arantes RL. Classification of cardiorespiratory fitness using the six-minute walk test in adults: Comparison with cardiopulmonary exercise testing. Pulmonology. 2021 Nov-Dec;27(6):500-508. doi: 10.1016/j.pulmoe.2021.03.006. Epub 2021 May 4. PMID 33958319
- [Background] Liu Y, Zhu J, Guo Z, Yu J, Zhang X, Ge H, Zhu Y. Estimated cardiorespiratory fitness and incident risk of cardiovascular disease in China. BMC Public Health. 2023 Nov 24;23(1):2338. doi: 10.1186/s12889-023-16864-5. PMID 38001416
- [Background] Lang JJ, Prince SA, Merucci K, Cadenas-Sanchez C, Chaput JP, Fraser BJ, Manyanga T, McGrath R, Ortega FB, Singh B, Tomkinson GR. Cardiorespiratory fitness is a strong and consistent predictor of morbidity and mortality among adults: an overview of meta-analyses representing over 20.9 million observations from 199 unique cohort studies. Br J Sports Med. 2024 May 2;58(10):556-566. doi: 10.1136/bjsports-2023-107849. PMID 38599681
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36646903/